CLINICAL TRIAL: NCT04939896
Title: Study on the Trajectories of Rehabilitation Compliance in Stroke Patients Based on Latent Growth Mixture Model
Brief Title: Study on the Trajectories of Rehabilitation Compliance in Stroke Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-1062
Record Dates: First submitted 2021-06-09; First posted 2021-06-25 (Actual); Last update posted 2021-06-25 (Actual); Status verified 2021-06

CONDITIONS: Stroke, Acute
Keywords: Rehabilitation; stroke; medical adherence; trajectory
MeSH Terms: conditions — Stroke | interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Compliance with rehabilitation: The patients' compliance with rehabilitation was followed up at 2, 6, 8, 12 and 24 weeks after onset, respectively
  Interventions: Other: observation

INTERVENTIONS:
Other: observation — Observed patients' compliance with rehabilitation at different time

SUMMARY:
To describe the general trajectories of rehabilitation compliance in first-onset stroke patients within 6 months, and to identify the heterogeneous development trajectory of different subgroups based on the mixed model of latent growth.To explore the predictors of different change tracks of rehabilitation compliance of stroke patients from the perspectives of biological, psychological and social factors, so as to provide the basis for formulating precise nursing intervention measures.

DETAILED DESCRIPTION:
To describe the general trajectories of rehabilitation compliance in first-onset stroke patients within 6 months. To recruit first-onset stroke patients undergoing rehabilitation and collect the general data. Telephone follow-up at 2 weeks, 6 weeks, 8 weeks, 12 weeks and 24 weeks after the onset. Based on the biological-psychosocial medical model and literature, biological, psychological and sociological factors were screened. The patient rehabilitation adherence level in different periods was measured. Latent Growth Mixture Model (LGMM) was used to investigate the general trend of rehabilitation compliance in patients with first-episode stroke within 6 months. Latent Class Growth Analysis (LCGA) method in Latent Growth hybrid model was used to identify the track of heterogeneous change. Multivariate Logistic regression analysis was used to explore the predictors of different subgroups of change trajectories relative to other subgroups.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with stroke by CT or MR;

  * Patients with first onset (within 14 days of onset); ③ limb dysfunction (muscle strength ≤4); ④ Age: ≥18 years old; ⑤ Awareness (NIHSS consciousness level ≤1 point);

    * Informed consent of patients.

Exclusion Criteria:

* Patients with deep vein thrombosis;

  * fracture patients;

    * a history of severe cardiopulmonary dysfunction and craniocerebral trauma;

      * recurrent stroke during the study; ⑤patients with severe mental disorders; ⑥ Mixed aphasia patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We recruited first-episode stroke patients who needed rehabilitation exercise in the Department of Neurology of a Grade A general hospital.After the approval of the ethics committee of the hospital, the purpose and process of the study were explained to the patients and their families, and the informed consent was signed.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-01-19 (Actual); Primary Completion 2022-02-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Motor Functional Exercise Compliance Scale for Stroke Patients | Week 2
  The full score is 56 points, and the higher the cumulative score of each item, the higher the level of compliance.
Motor Functional Exercise Compliance Scale for Stroke Patients | Week 6
  The full score is 56 points, and the higher the cumulative score of each item, the higher the level of compliance.
Motor Functional Exercise Compliance Scale for Stroke Patients | Week 8
  The full score is 56 points, and the higher the cumulative score of each item, the higher the level of compliance.
Motor Functional Exercise Compliance Scale for Stroke Patients | Week 12
  The full score is 56 points, and the higher the cumulative score of each item, the higher the level of compliance.
Motor Functional Exercise Compliance Scale for Stroke Patients | Week 24
  The full score is 56 points, and the higher the cumulative score of each item, the higher the level of compliance.

CONTACTS AND LOCATIONS:
Overall Officials: Yuping Yuping, master, Principal Investigator — Nursing Department Second Affiliated Hospital of Zhejiang University School of Medicine
Locations (1):
- Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No